CLINICAL TRIAL: NCT02351167
Title: Genetically Informed Smoking Cessation Trial
Acronym: GISC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201305128; 1R01DA038076-01A1 (NIH)
Record Dates: First submitted 2015-01-26; First posted 2015-01-30 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Counseling; Genetics and Genomics
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine; Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combination NRT and Counseling (Active Comparator): Combination Nicotine replacement therapy (cNRT) (patch and lozenge) and smoking cessation counseling will be provided to participants. Lozenges will be given for 12 weeks with a 1 week pre-quit titration and patch for 12 weeks. Seven smoking counseling sessions will be given during treatment.
  Interventions: Drug: Combination NRT (Nicotine patch, Nicotine lozenge); Behavioral: Intensive smoking counseling
- Varenicline (Chantix) and Counseling (Active Comparator): Varenicline (pill) and smoking cessation counseling will be provided to participants for 12 weeks with 1 week pre-quit titration. Seven smoking cessation counseling sessions will be given during treatment.
  Interventions: Drug: Varenicline; Behavioral: Intensive smoking counseling
- Placebo Medicine and Counseling (Placebo Comparator): Placebo pill and smoking cessation counseling will be provided to participants for 12 weeks with 1 week pre-quit titration. Placebo lozenges will be given for 12 weeks with a 1 week pre-quit titration and patch for 12 weeks. Seven smoking counseling sessions will be given during treatment.
  Interventions: Drug: Placebo; Behavioral: Intensive smoking counseling

INTERVENTIONS:
Drug: Combination NRT (Nicotine patch, Nicotine lozenge)
  Other Names: Nicoderm CQ; Nicotine Polacrilex Lozenge
  Arms: Combination NRT and Counseling
Drug: Varenicline
  Other Names: Chantix
  Arms: Varenicline (Chantix) and Counseling
Drug: Placebo
  Arms: Placebo Medicine and Counseling
Behavioral: Intensive smoking counseling

SUMMARY:
The investigators' goal is to identify the most appropriate smoking cessation treatments for smokers based on genetic information. Smokers try to quit smoking but relapses are common.

DETAILED DESCRIPTION:
The investigators' goal is to determine whether genetic markers can be used to optimize smoking cessation pharmacotherapy to enhance efficacy, medication adherence, and reduce side effects. Smoking is a leading cause of preventable death and disability, and smoking cessation reverses the risk of mortality. However, cessation failure is common despite available cessation medications, which are associated with different efficacy, side effects, adherence, use constraints, and costs. This challenge can be addressed by improving current treatments via personalized medicine based on individual genetic markers to maximize efficacy and minimize side effects.

The investigators propose a prospective, genotype-based stratified randomization trial to compare two smoking cessation medications (combination NRT [patch and lozenge], varenicline vs. placebo) for 3 months in 720 smokers with known genotypes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥21 years of age), seeking treatment for smoking cessation.
2. Able to speak English,
3. Active smoking (Cigarettes Per Day (CPD) ≥5), and exhaled Carbon Monoxide (CO) ≥8 ppm
4. Agree to participate in this randomized smoking cessation trial with follow up assessments up to 12 months.

Exclusion Criteria:

1. Pregnancy or breast feeding,
2. Active use or recent use (< or equal to 1 month) of medication or e-cigarettes for nicotine dependence/smoking cessation, or use of e-cigarettes for more than 9 days in the prior month,
3. Allergy to nicotine patch, lozenge, or varenicline,
4. Unwillingness to prevent pregnancy during the medication phase and 1 month afterwards (women only),
5. Significant cardiac conditions (myocardial infarction, unstable angina, coronary angioplasty, cardiac bypass) or serious arrhythmia in past 6 months,
6. Current heavy alcohol consumption (≥6 drinks/day, 6 days/week),
7. Active psychosis or poorly controlled depression within the past 6 months,
8. Any prior suicide attempt or suicidal ideation within the past 6 months,
9. End stage renal disease with hemodialysis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Shiun Chen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen LS, Baker TB, Miller JP, Bray M, Smock N, Chen J, Stoneking F, Culverhouse RC, Saccone NL, Amos CI, Carney RM, Jorenby DE, Bierut LJ. Genetic Variant in CHRNA5 and Response to Varenicline and Combination Nicotine Replacement in a Randomized Placebo-Controlled Trial. Clin Pharmacol Ther. 2020 Dec;108(6):1315-1325. doi: 10.1002/cpt.1971. Epub 2020 Aug 4. PMID 32602170
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 05/20/2015 and closed to participant enrollment on 07/23/2018.
Pre-assignment Details: -The study consented 894 participants and 72 were excluded after consenting due to no longer wanting to participate or not meeting all the eligibility criteria prior to randomization. The 72 were not considered enrolled in the study per the policy of the institution.
Period: Overall Study
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling
Started | 275 | 274 | 273
Completed | 256 | 256 | 252
Not Completed | 19 | 18 | 21
Not completed — Withdrawal by Subject | 19 | 18 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling | Total
Number analyzed (Participants) | 275 | 274 | 273 | 822
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 261 | 262 | 258 | 781
  >=65 years | 14 | 12 | 15 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.2) | 46.6 (11.0) | 46.6 (11.5) | 46.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 144 | 161 | 449
  Male | 131 | 130 | 112 | 373
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 5 | 18
  Not Hispanic or Latino | 271 | 265 | 268 | 804
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 97 | 91 | 82 | 270
  White | 168 | 169 | 179 | 516
  More than one race | 5 | 4 | 9 | 18
  Unknown or Not Reported | 2 | 8 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 275 | 274 | 273 | 822

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Quit Rate
Description: The definition of this measure requires: (a) no self-reported smoking (not even a puff of a cigarette) for at least the 7 days prior to the assessment, and (b) biochemical verification of abstinence.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling
Number analyzed (Participants) | 275 | 274 | 273
Participants | 55 | 70 | 24

2. Secondary Outcome: Continuous Abstinence
Description: The definition of this measure requires: Not taking even 1 cigarette puff from target quit date to end of treatment.
Time Frame: 12 weeks (with first 1 week initial grace period)
Measure: Count of Participants; unit: Participants
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling
Number analyzed (Participants) | 275 | 274 | 273
Participants | 43 | 46 | 21

3. Secondary Outcome: 7-day Point Prevalence Quit Rate
Description: as for outcome 1
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling
Number analyzed (Participants) | 275 | 274 | 273
Participants | 37 | 56 | 25

4. Secondary Outcome: Number of Days to Lapse
Description: * The number of days to lapse is defined as the number of days from the target quit date until the participant reports smoking (even a single puff).
  * Participants who did not lapse by the end of the 52 weeks and participants who had missing information on lapse are not included in the overall number of participants analyzed
Time Frame: Assessed from the target quit day through 52 weeks
Population: 26 participants in Combination NRT & Counseling, 19 participants in Varenicline (Chantix) & Counseling, & 16 participants in Placebo Medicine & Counseling did not lapse by the end of the 52 weeks. 4 participants in Combination NRT & Counseling, 9 participants in Varenicline (Chantix) & Counseling, & 5 participants had missing information on lapse.
Measure: Mean (Standard Error); unit: days
Groups:
- 3 Arms Combined: This is the total of all participants who were enrolled in all 3 arms including Combination NRT and Counseling, Varenicline (Chantix) and Counseling, and Placebo Medicine and Counseling.
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling | 3 Arms Combined
Number analyzed (Participants) | 245 | 246 | 252 | 743
days | 16.78 (2.48) | 20.47 (3.22) | 11.85 (2.07) | 16.33 (1.52)

5. Secondary Outcome: Number of Days to Relapse
Description: * The number of days to relapse is defined as the number of days from the target quit day until the first of seven consecutive days of smoking.
  * Participants who did not relapse by the end of the 52 weeks and participants who had missing information on relapse are not included in the overall number of participants analyzed
Time Frame: Assessed from the target quit day through 52 weeks
Population: 76 participants in Combination NRT & Counseling, 66 participants in Varenicline (Chantix) & Counseling, & 51 participants in Placebo Medicine & Counseling did not relapse by the end of 52 weeks. 4 participants in Combination NRT & Counseling, 9 participants in Varenicline (Chantix) & Counseling, & 5 participants had missing information on relapse
Measure: Mean (Standard Error); unit: days
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling | 3 Arms Combined
Number analyzed (Participants) | 195 | 199 | 217 | 611
days | 44.83 (4.25) | 45.01 (5.04) | 28.87 (3.75) | 39.22 (2.53)

6. Secondary Outcome: Initial Cessation
Description: Defined as at least 1 day of abstinence during the first 7 days after the target quit day.
Time Frame: Assessed for the first seven days after the target quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling
Number analyzed (Participants) | 275 | 274 | 273
Participants | 217 | 186 | 172

7. Secondary Outcome: Longitudinal Models of Abstinence Outcomes Across Multiple Time Points
Description: -The definition of this measure requires; no self-reported smoking (not even a puff of a cigarette) for at least 7 days prior to the assessment.
Time Frame: 0-52 Weeks
Population: Participants who had missing data are not included in the number of participants analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling | 3 Arms Combined
Number analyzed (Participants) | 271 | 268 | 270 | 809
Participants
  0 weeks - Abstinence | 5 | 3 | 0 | 8
  1 week - Abstinence: number analyzed (Participants) | 266 | 263 | 260 | 789
  1 week - Abstinence | 91 | 94 | 70 | 255
  2 week - Abstinence: number analyzed (Participants) | 260 | 258 | 258 | 776
  2 week - Abstinence | 119 | 105 | 70 | 294
  4 week - Abstinence: number analyzed (Participants) | 251 | 253 | 248 | 752
  4 week - Abstinence | 112 | 114 | 74 | 300
  12 week - Abstinence: number analyzed (Participants) | 248 | 252 | 238 | 738
  12 week - Abstinence | 81 | 88 | 49 | 218
  26 week - Abstinence: number analyzed (Participants) | 244 | 242 | 240 | 726
  26 week - Abstinence | 75 | 82 | 49 | 206
  52 week - Abstinence: number analyzed (Participants) | 234 | 244 | 226 | 704
  52 week - Abstinence | 68 | 77 | 43 | 188

8. Secondary Outcome: Longitudinal Models of Smoking Quantity in Cigarettes Per Day Outcomes Across Multiple Time Points.
Description: The definition of this measure requires self-reported cigarettes per day.
Time Frame: 0-52 Weeks
Population: Participants who had missing data are not included in the number of participants analyzed
Measure: Mean (Standard Error); unit: cigarettes per day
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling | 3 Arms Combined
Number analyzed (Participants) | 265 | 262 | 261 | 788
cigarettes per day
  0 week | 2.50 (0.38) | 2.95 (0.32) | 3.74 (0.38) | 3.06 (0.21)
  1 week: number analyzed (Participants) | 265 | 261 | 258 | 784
  1 week | 3.06 (0.40) | 3.18 (0.34) | 4.46 (0.37) | 3.56 (0.22)
  2 week: number analyzed (Participants) | 257 | 257 | 254 | 768
  2 week | 3.43 (0.39) | 3.08 (0.35) | 5.00 (0.41) | 3.83 (0.22)
  4 week: number analyzed (Participants) | 249 | 251 | 247 | 747
  4 week | 4.08 (0.43) | 3.63 (0.41) | 5.79 (0.43) | 4.49 (0.25)
  12 week: number analyzed (Participants) | 240 | 245 | 238 | 723
  12 week | 6.38 (0.53) | 5.75 (0.50) | 8.33 (0.52) | 3.50 (0.30)
  26 week: number analyzed (Participants) | 233 | 241 | 226 | 700
  26 week | 7.68 (0.58) | 7.09 (0.53) | 9.38 (0.57) | 8.03 (0.32)
  52 week: number analyzed (Participants) | 225 | 240 | 219 | 684
  52 week | 7.67 (0.59) | 7.76 (0.57) | 8.98 (0.55) | 8.12 (0.33)

9. Secondary Outcome: Medication Adherence
Description: Adherence is the proportion of expected medication (varenicline, patch, lozenge) taken as advised during pre-quit week to week 12
Time Frame: Pre-quit week to Week 12
Population: Not all participants were evaluable for this outcome measure due to data not being available. Also the Varenicline (Chantix) and Counseling Arm did not receive the lozenge or the patch. The Combination NRT and Counseling Arm did not receive Varenicline (Chantix)
Measure: Mean (Standard Deviation); unit: proportion of expected medication taken
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling
Number analyzed (Participants) | 234 | 242 | 233
proportion of expected medication taken
  Patch: number analyzed (Participants) | 234 | 0 | 233
  Patch | 0.65 (0.34) |  | 0.57 (0.36)
  Lozenge: number analyzed (Participants) | 234 | 0 | 233
  Lozenge | 0.57 (0.39) |  | 0.57 (0.38)
  Varenicline (Chantix): number analyzed (Participants) | 0 | 242 | 233
  Varenicline (Chantix) |  | 0.67 (0.32) | 0.70 (0.35)

10. Secondary Outcome: Side Effects
Description: All reported side effects (occurring>4%) will be summarized and presented for the study. In addition, the investigators will further identify a pre-specified set of key side effects as being related to drug agonist effects (e.g., nausea, vomiting, racing heart, headache, and sleep disturbance). These will be analyzed as rate of occurrence during the period of medication use.
Time Frame: Pre-quit week to Week 12
Population: Not all participants were evaluable for this outcome measure due to data not being available.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling
Number analyzed (Participants) | 229 | 241 | 208
Participants
  Nausea | 53 | 92 | 59
  Vomiting | 28 | 36 | 27
  Racing Heart | 27 | 24 | 17
  Headache | 81 | 81 | 71
  Sleep Disturbance | 49 | 55 | 42

11. Secondary Outcome: Withdrawal
Description: * Withdrawal severity is assessed by Wisconsin Smoking Withdrawal Scale (WSWS), there are 28 items.
  * Participants rate each item on a scale of 0-4 (0=Strongly disagree, 1=Disagree, 2=Feel neutral, 3=Agree, 4=Strongly agree). The subscale to each item is determined on how high they agree on the scale. For some items, the subscale is determined on how low they agreed. Each score is determined by the mean of each item that applies. Higher means indicate greater withdrawal.
  * The scores were calculated by averaging a mean score of each item for each participant with data from time point pre-quit, quit, week 1, week 2, and week 4. The mean score for each participant was averaged for each item and a mean score was taken for each treatment condition (cNRT, Varenicline, Placebo). These data are reported as mean withdrawal scores and not change in withdrawal scores.
Time Frame: Pre-quit, quit, week 1, week 2, and week 4
Population: Not all participants were evaluable for this outcome measure due to data not being available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling
Number analyzed (Participants) | 261 | 263 | 253
score on a scale
  Anger | 1.33 (0.75) | 1.49 (0.81) | 1.47 (.79)
  Anxiety | 1.69 (0.79) | 1.81 (0.90) | 1.82 (0.83)
  Concentration | 1.28 (0.64) | 1.48 (0.76) | 1.42 (0.76)
  Craving | 2.29 (0.85) | 2.20 (0.86) | 2.50 (0.83)
  Hunger | 2.11 (0.84) | 2.28 (0.80) | 2.17 (0.79)
  Sadness | 1.01 (0.63) | 1.11 (0.69) | 1.11 (0.61)
  Sleep | 1.49 (0.82) | 1.70 (0.89) | 1.54 (0.92)

ADVERSE EVENTS:
Time Frame: Adverse events were collected until from enrollment until 1 year post target quit date. Post-study adverse events will be recorded when the subject volunteers to report such events to the investigator team.
Description: Adverse events are assessed in each follow-up visit to the end of the trial. With respect to the pharmacotherapy, participants will be made aware of the common side effects before they consent to participate in the study. During each study visit, participants are asked about common side effects associated with the drug(s) as well as any other symptoms participants report regardless of attribution to the drug(s).
Arm/Group | Combination NRT and Counseling | Varenicline (Chantix) and Counseling | Placebo Medicine and Counseling
All-Cause Mortality (participants affected / at risk) | 3/275 | 2/274 | 4/273
Serious Adverse Events (participants affected / at risk) | 23/275 | 17/274 | 27/273
Other Adverse Events (participants affected / at risk) | 193/275 | 204/274 | 175/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination NRT and Counseling (N=275) | Varenicline (Chantix) and Counseling (N=274) | Placebo Medicine and Counseling (N=273)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Death due to cardiorespiratory arrest (Cardiac disorders) | 1 | 0 | 0
Death due to congestive heart failure (Cardiac disorders) | 0 | 0 | 1
Heart failure (Cardiac disorders) | 0 | 0 | 1
Left bundle branch block (Cardiac disorders) | 1 | 0 | 0
Death due to diabetic coma (Endocrine disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Type 2 Diabetes (Endocrine disorders) | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulosis (Gastrointestinal disorders) | 0 | 2 | 0
Hemorrhoid (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Death, unknown (General disorders) | 0 | 1 | 0
Death due to natural causes (General disorders) | 1 | 0 | 0
Ammonia poisoning of liver (Hepatobiliary disorders) | 1 | 0 | 0
Antibiotic spacer for MRSA infection in knee (Infections and infestations) | 0 | 1 | 0
Cellulitis, right hand (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Surgical incision site infection (post-surgery) (Infections and infestations) | 0 | 0 | 1
Infection of second toe on left foot (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
MRSA infection in knee (Infections and infestations) | 0 | 1 | 0
Malaria (Infections and infestations) | 0 | 0 | 1
Severe sinus infection (Infections and infestations) | 1 | 0 | 0
Severe tooth infection (Infections and infestations) | 0 | 0 | 1
Broken arm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Broken collarbone (Injury, poisoning and procedural complications) | 1 | 0 | 0
Broken ribs (Injury, poisoning and procedural complications) | 1 | 0 | 1
Cervical disc fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Complication from gastric bypass surgery (Injury, poisoning and procedural complications) | 0 | 0 | 1
Death due to heroin overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gunshot wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Homicide by gunshot (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Motor vehicle accident (injury of intervertebral discs T10-12) (Injury, poisoning and procedural complications) | 0 | 1 | 0
Partial amputation of leg due to MRSA infection (Injury, poisoning and procedural complications) | 0 | 1 | 0
Struck by vehicle (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sternum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Inter-vertebral dis herniation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Death due to Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Death due to brain tumor complications (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung cancer (stage 4) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bell's palsy (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 1 | 1
Alcohol dependence (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Bipolar depression (Psychiatric disorders) | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 1
Unspecified mood disorder (Psychiatric disorders) | 0 | 1 | 0
Death due to kidney failure (Renal and urinary disorders) | 0 | 0 | 1
Kidney stone (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Stage 4 endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0
Asthmatic episode (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Chronic sinus necrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Thoracic outlet syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Trouble breathing due to COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Abdominal hysterectomy due to endometriosis (Surgical and medical procedures) | 0 | 1 | 0
Foot surgery to fix broken toes on right foot (Surgical and medical procedures) | 1 | 0 | 0
Hip replacement surgery (Surgical and medical procedures) | 2 | 0 | 1
Hysterectomy due to cervical cancer (Surgical and medical procedures) | 0 | 1 | 0
Hysterectomy due to enlarged fallopian tubes (Surgical and medical procedures) | 1 | 0 | 0
Knee surgery for osteoarthritis (Surgical and medical procedures) | 0 | 0 | 1
Left knee replacement (Surgical and medical procedures) | 1 | 0 | 0
Minor procedure to clean wound on right foot (Surgical and medical procedures) | 1 | 0 | 0
Surgery for aortic valve stenosis and cardiac bypass (Surgical and medical procedures) | 0 | 0 | 1
Urethral sling surgery due to urinary incontinence (Surgical and medical procedures) | 0 | 1 | 0
Abdominal aortic aneurysm (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Pulmonary embolism (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination NRT and Counseling (N=275) | Varenicline (Chantix) and Counseling (N=274) | Placebo Medicine and Counseling (N=273)
Nausea (Gastrointestinal disorders) | 53 | 92 | 59
Vomiting (Gastrointestinal disorders) | 28 | 36 | 27
Headache (Nervous system disorders) | 81 | 81 | 71
Rapid, slow, pounding, or irregular heartbeat (Cardiac disorders) | 27 | 24 | 17
Insomnia (Psychiatric disorders) | 49 | 55 | 42
Vivid dreams (Psychiatric disorders) | 63 | 100 | 60
Dizziness (Nervous system disorders) | 41 | 52 | 39
Weakness (General disorders) | 25 | 32 | 32
Sweating (Skin and subcutaneous tissue disorders) | 46 | 40 | 29
Itching/hives (Skin and subcutaneous tissue disorders) | 35 | 29 | 16
Rash (Skin and subcutaneous tissue disorders) | 33 | 18 | 22
Swelling in face or hands (Immune system disorders) | 15 | 10 | 16
Swelling or tingling in mouth or throat (Immune system disorders) | 20 | 8 | 12
Mouth problems (e.g. pain or sore) (Gastrointestinal disorders) | 21 | 20 | 21
Indigestion (Gastrointestinal disorders) | 41 | 51 | 36
Hiccups (Respiratory, thoracic and mediastinal disorders) | 34 | 43 | 22
Chest tightness (Cardiac disorders) | 24 | 24 | 16
Trouble breathing (Respiratory, thoracic and mediastinal disorders) | 16 | 21 | 22
Feeling worried, nervous, scared, or anxious (Psychiatric disorders) | 50 | 64 | 58
Feeling panicky or having panic attacks (Psychiatric disorders) | 22 | 23 | 22
Feeling agitated and restless (Psychiatric disorders) | 47 | 56 | 43
Feeling hostile or angry towards others (Psychiatric disorders) | 15 | 32 | 23
Feeling significantly down, depressed, or hopeless (Psychiatric disorders) | 47 | 58 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT02351167/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT02351167/ICF_001.pdf